CLINICAL TRIAL: NCT03808805
Title: Aprepitant Versus Hydroxyzine in Association With Cytoreductive Treatments for Patients With Myeloproliferative Neoplasia Suffering From Persistent Aquagenic Pruritus.
Brief Title: Aprepitant Versus Hydroxyzine in Persistent Aquagenic Pruritus for Patients With Myeloproliferative Neoplasms
Acronym: APHYPAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ApHyPAP 29BRC18.0036; 2018-000426-66 (EudraCT Number)
Record Dates: First submitted 2018-09-26; First posted 2019-01-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2024-08

CONDITIONS: Myeloproliferative Disorder; Aquagenic Pruritus
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Aprepitant; Hydroxyzine

STUDY DESIGN:
Intervention Model Description: Phase 3, randomized prospective study, double blind-double placebo
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- studied group (Experimental): Aprepitant 80 mg daily - 14 days Plus placebo of Hydroxyzine - 14 days
  Interventions: Drug: Aprepitant 80 mg; Drug: Placebo of Hydroxyzine
- comparative group (Active Comparator): Hydroxyzine 25 mg/d - 14 days Plus placebo of Aprepitant - 14 days
  Interventions: Drug: Hydroxyzine 25mg; Drug: Placebo of Aprepitant

INTERVENTIONS:
Drug: Aprepitant 80 mg — oral therapy - daily dose - 14 days
  Arms: studied group
Drug: Hydroxyzine 25mg — oral therapy - daily dose - 14 days
  Arms: comparative group
Drug: Placebo of Hydroxyzine — oral therapy - daily dose - 14 days
  Arms: studied group
Drug: Placebo of Aprepitant — oral therapy - daily dose - 14 days
  Arms: comparative group

SUMMARY:
Phase 3, randomized prospective study, double blind-double placebo, testing oral therapies APREPITANT versus HYDROXYZINE in patients followed for myeloproliferative neoplasms and suffering of persistent aquagenic pruritus.

DETAILED DESCRIPTION:
Identification of patients with myeloproliferative neoplasms and aquagenic pruritus. Evaluation of the intensity of the aquagenic pruritus. Patients with value >5/10 on the VAS (Visual Analogue Scale ) are proposed to participate to the protocole. Randomization between the two treatments. Duration of the treatment : 14 days. Regular evaluation of efficacity of the drugs (questionnaires). Evaluations will stop 2 months after the last intake. Blood samples will be collected before and after the intakes to study cytokine and neuropeptide levels.

ELIGIBILITY:
Inclusion Criteria:

* Major patients with myeloproliferative neoplasms (polycythemia vera, essential thrombocythaemia or myelofibrosis)
* and treated with hydroxyurea, pipobroman, anagrelide, α2a pegylated interferon, ruxolitinib or bled for more than 6 months
* and suffering of persistent aquagenic pruritus
* and with a pruritus intensity on Analogic Visual Scale >5/10
* patients who gave their written consent for participation in the study

Exclusion Criteria:

* patients with a physical or psychological disability to sign the consent form
* patients with myeloproliferative neoplasms and suffering of aquagenic pruritus but only treated by aspirin
* patients already included in another therapeutic protocol
* patients with diffuse dermatological disease where pruritus may be present (psoriasis, atopic dermatitis, prurigo
* patients already on anti-anxiety and / or anti-depressant treatment
* patients with absolute contraindications to the use of Aprepitant or Hydroxyzine
* hypersensitivity to Aprepitant and / or Hydroxyzine or to any of their excipients
* lactose intolerance
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Reduction of pruritus intensity below (or equal) 3/10 on the VAS (Visual Analogue Scale ) | at 15 days
  number of patients with a pruritus intensity below (or equal) 3/10 on the VAS (Visual Analogue Scale wich measure the intensity of symptoms of pruritus, 0 is minimum and 10 is maximum intensity of symptoms)

SECONDARY OUTCOMES:
Reduction of pruritus intensity below (or equal) 3/10 on the VAS (Visual Analogue Scale ) | at 60 days
  number of patients with a pruritus intensity below (or equal) 3/10 on the VAS (Visual Analogue Scale wich measure the intensity of symptoms of pruritus, 0 is minimum and 10 is maximum intensity of symptoms)
Cessation of pruritus | at 15 days
  number of patients with a pruritus intensity at 0/10 on the VAS (Visual Analogue Scale wich measure the intensity of symptoms of pruritus, 0 is minimum and 10 is maximum intensity of symptoms) )
Cessation of pruritus | at 60 days
  number of patients with a pruritus intensity at 0/10 on the VAS (Visual Analogue Scale wich measure the intensity of symptoms of pruritus, 0 is minimum and 10 is maximum intensity of symptoms))
Time observed to decreased the VAS to 3/10 | 01 to 60 days
  number of days to obtain an intensity of pruritus at 3/10 on the VAS (Visual Analogue Scale )
Duration of treatment effectiveness | 1 to 60 days
  number of days the VAS (Visual Analogue Scale ) is below (or equal) 3/10
Adverse event occurring during the association therapeutic | at 15 days
  type of adverse event occuring during the treatment period
Number of prematurely discontinued anti-pruritic treatment | at 15 days
  Total number of prematurely discontinued treatments for all subjects
Complete blood count (normal or abnormal) | 1 to 60 days
  number of patients with hematologic remission : hematocrit <45% with leukocytes <10 giga/l and platelets <400 giga/l
Quality of life through the use of validated questionnaire : the MPN-SAF (Myeloproliferative Neoplasm Symptom Assessment Form) questionnaire | at J0 (day of inclusion)
  Evaluation of quality of life by completion of the MPN-SAF (Myeloproliferative Neoplasm Symptom Assessment Form calculated as the mean score for 10 items. Questions focus on fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers) questionnaire
Quality of life through the use of validated questionnaire : the PASYMPLE questionnaire | at J0 (day of inclusion)
  Evaluation of quality of life by completion of the PASYMPLE (evaluation of pruritus with 7 questions about occurence, timing, intensity and localisation of pruritus) questionnaire
Quality of life through the use of validated questionnaire : the MPN-SAF (Myeloproliferative Neoplasm Symptom Assessment Form) questionnaire | at 15 days
  Evaluation of quality of life by completion of the MPN-SAF (Myeloproliferative Neoplasm Symptom Assessment Form calculated as the mean score for 10 items. Questions focus on fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers)questionnaire
Quality of life through the use of validated questionnaire : the PASYMPLE questionnaire | at 15 days
  Evaluation of quality of life by completion of the PASYMPLE (evaluation of pruritus with 7 questions about occurence, timing, intensity and localisation of pruritus) questionnaire
Quality of life through the use of validated questionnaires : the MPN-SAF (Myeloproliferative Neoplasm Symptom Assessment Form) questionnaire | at 30 days
  Evaluation of quality of life by completion of the MPN-SAF (Myeloproliferative Neoplasm Symptom Assessment Form calculated as the mean score for 10 items. Questions focus on fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers) questionnaire
Quality of life through the use of validated questionnaire : the PASYMPLE questionnaire | at 30 days
  Evaluation of quality of life by completion of the PASYMPLE (evaluation of pruritus with 7 questions about occurence, timing, intensity and localisation of pruritus) questionnaire
Quality of life through the use of validated questionnaire : the MPN-SAF (Myeloproliferative Neoplasm Symptom Assessment Form) questionnaire | at 45 days
  Evaluation of quality of life by completion of the MPN-SAF(Myeloproliferative Neoplasm Symptom Assessment Form calculated as the mean score for 10 items. Questions focus on fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers) questionnaire
Quality of life through the use of validated questionnaire : the PASYMPLE questionnaire | at 45 days
  Evaluation of quality of life by completion of the PASYMPLE (evaluation of pruritus with 7 questions about occurence, timing, intensity and localisation of pruritus) questionnaire
Quality of life through the use of validated questionnaire : the MPN-SAF (Myeloproliferative Neoplasm Symptom Assessment Form) questionnaire | at 60 days
  Evaluation of quality of life by completion of the MPN-SAF (Myeloproliferative Neoplasm Symptom Assessment Form calculated as the mean score for 10 items. Questions focus on fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers) questionnaire
Quality of life through the use of validated questionnaire : the PASYMPLE questionnaire | at 60 days
  Evaluation of quality of life by completion of the PASYMPLE (evaluation of pruritus with 7 questions about occurence, timing, intensity and localisation of pruritus) questionnaire
Quantification of the change of plasma concentrations of cytokines and neuropeptides | at J0 (day of inclusion)
  Plasma concentrations of cytokines (ng/L) and neuropeptides (ng/mL)
Quantification of the change of plasma concentrations of cytokines and neuropeptides | at 15 days
  Plasma concentrations of cytokines (ng/L) and neuropeptides (ng/mL)
Quantification of the change of plasma concentrations of cytokines and neuropeptides | at 30 days
  Plasma concentrations of cytokines (ng/L) and neuropeptides (ng/mL)
Quantification of the change of plasma concentrations of cytokines and neuropeptides | at 60 days
  Plasma concentrations of cytokines (ng/L) and neuropeptides (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe IANOTTO, MD, PhD, Principal Investigator — Hématologie Clinique-Institut de Cancéro-Hématologie
Locations (11):
- France (11):
  - CHRU de Brest - Hôpital Morvan, Brest, Brest Cedex
  - Centre Hospitalier de Cornouaille, Quimper, Quimper
  - CHU d'Angers, Angers
  - CHU de Caen, Caen
  - Centre Hospitalier de Douarnenez, Douarnenez
  - CHU Grenoble Alpes, Grenoble
  - Centre Léon Bérard, Lyon
  - Centre Hospitalier des Pays de Morlaix, Morlaix
  - CHU de Nantes, Nantes
  - Hôpital Pontchaillou, Rennes
  - Hôpital Yves Le Foll, Saint-Brieuc

REFERENCES:
- [Derived] Le Gall-Ianotto C, Verdet R, Nowak E, Le Roux L, Gasse A, Fiedler A, Carlhant-Kowalski D, Marcorelles P, Misery L, Ianotto JC. Rationale and design of the multicentric, double-blind, double-placebo, randomized trial APrepitant versus HYdroxyzine in association with cytoreductive treatments for patients with myeloproliferative neoplasia suffering from Persistent Aquagenic Pruritus. Trial acronym: APHYPAP. Trials. 2021 Dec 19;22(1):938. doi: 10.1186/s13063-021-05864-8. PMID 34923994